CLINICAL TRIAL: NCT07156552
Title: Effectiveness of Protein SupplementatIon Combined With Resistance Exercise Training to Counteract Disproportional Fat-Free Mass Loss Following Metabolic-Bariatric Surgery: The ENRICHED Study
Brief Title: Protein Supplementation and Resistance Training to Prevent Fat-Free Mass Loss Following Metabolic-Bariatric Surgery
Acronym: ENRICHED
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Amsterdam University Medical Centers (UMC), Location Academic Medical Center (AMC) (Other); ZonMw: The Netherlands Organisation for Health Research and Development (Other); Nederlandse Obesitas Kliniek (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NL87367.091.24
Record Dates: First submitted 2025-07-22; First posted 2025-09-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-06

CONDITIONS: Bariatric Surgery; Fat Free Mass
Keywords: Metabolic-Bariatric Surgery; Bariatric Surgery; Sleeve Gastrectomy; Roux-en Y Gastric Bypass; Protein Supplementation; Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group - Standard care (No Intervention)
- Intervention group - Enriched care (Experimental)
  Interventions: Behavioral: Resistance exercise training and protein supplementation

INTERVENTIONS:
Behavioral: Resistance exercise training and protein supplementation — The intervention consists of two components:
  1. Resistance Exercise Training Participants will engage in a 24-week resistance training program. This program includes one supervised session per week supervised by a qualified kinesiologist, complemented by two to three additional unsupervised sessions per week performed at home.
  2. Protein Supplementation
  Participants will receive daily protein supplements for a total duration of 12 weeks. The dosage will be progressively increased:
  * 20 grams per day during weeks 1-4
  * 40 grams per day during weeks 5-8
  * 60 grams per day during weeks 9-12 After the 12-week supplementation period, participants will receive additional dietary counseling sessions with a dietitian. These sessions aim to support the maintenance of adequate protein intake through dietary intake.
  Arms: Intervention group - Enriched care

SUMMARY:
The goal of this clinical trial is to investigate the effects of daily protein supplementation and participation in a weekly supervised resistance training program on the prevention of excessive muscle mass loss following bariatric surgery. Patients treated at one of the participating centers will be invited to participate and will be randomly assigned to one of two groups.

Participants in group 1 will receive standard postoperative care as currently provided. Participants in group 2 will also receive standard care, but in addition, they will be asked to consume extra protein daily and take part in a supervised resistance training session once a week.

Previous research has shown that approximately one in five patients undergoing bariatric surgery experiences excessive muscle loss after the surgery. It is known that resistance training and protein intake can help maintain and even improve muscle mass. However, limited research has been conducted on the combined effects of protein supplementation and resistance training in patients after bariatric surgery. Therefore, the aim of this trial is to determine whether participants receiving the additional intervention experience less muscle mass loss compared to those receiving standard care alone.

ELIGIBILITY:
Inclusion Criteria:

* A scheduled metabolic-bariatric surgery (i.e. RYGB or Sleeve Gastrectomy)
* Participation in the NOK care program
* Able to understand and perform the study procedures

Exclusion Criteria:

* Allergic or sensitive for milk proteins, or lactose intolerant
* Diagnosed renal insufficiency
* Diagnosed intestinal diseases influencing the uptake of protein (i.e. active inflammatory bowel disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-06-20 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Prevalence of Fat-free mass loss/Total weight loss >30% | From enrollment to 3 months post-surgery

SECONDARY OUTCOMES:
Weight (kg) | From enrollment to 12 months post-surgery
Body Mass Index (kg/m2) | From enrollment to 12 months post-surgery
Body composition (fat-mass/fat-free mass) (kg) | From enrollment to 12 months post-surgery
Waist circumference (cm) | From enrollment to 12 months post-surgery
Blood pressure (mmHg) | From enrollment to 12 months post-surgery
Quadriceps isometric strength (kg) | From enrollment to 12 months post-surgery
Quadriceps isometric power (Watt) | From enrollment to 12 months post-surgery
Handgrip strength (kg) | From enrollment to 12 months post-surgery
Short Physical Performance Battery (SPPB) score (scale 1-12 points) | From enrollment to 12 months post-surgery
  Based on a balance test (0-4 points), a gait speed test (0-4 points), and a repeated chair stand (0-4 points)
VO2max (L/min) | From enrollment to 12 months post-surgery
  Assessment using the Astrand-Rhyming six minute cycle ergometer test
Incidence of gastrointestinal symptoms | From enrollment to 12 months post-surgery
  Assessment using the Gastrointestinal Symptom Rating Scale (GSRS) questionnaire
Difference in Health-Related Quality of Life (HRQoL) | From enrollment to 12 months post-surgery
  Assessment using the BODY-Q questionnaire
Healthcare consumption (costs) | From enrollment to 12 months post-surgery
Blood marker HOMA-IR | From enrollment to 12 months post-surgery
  Based on fasted insulin (microU/mL) and glucose (mmol/L) levels
Blood marker high-sensitivity C-Reactive Protein (hs-CRP) (mg/L) | From enrollment to 12 months post-surgery
Blood marker lipid profile | From enrollment to 12 months post-surgery
  Based on HDL-cholesterol (mg/dL), LDL-cholesterol (mg/dL), and triglycerides (mg/dL)

CONTACTS AND LOCATIONS:
Overall Officials: M. T.E. Hopman, Prof. Dr., Principal Investigator — Radboud University Medical Center
Locations (2):
- Netherlands (2):
  - Nederlandse Obesitas Kliniek, Amsterdam
  - Nederlandse Obesitas Kliniek, Nieuwegein

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] de Roos BM, Yeh LY, van den Hooff PS, Nuijten MAH, Twisk JWR, Liem RSL, van Acker GJD, Severens JL, Kambic T, Serlie MJM, Monpellier VM, Eijsvogels TMH, Hopman MTE, Karregat JHM. Effectiveness of protein supplementation combined with resistance training to counteract disproportional fat-free mass loss following metabolic bariatric surgery: rationale and design of the ENRICHED randomised controlled trial. BMJ Open. 2025 Dec 29;15(12):e108346. doi: 10.1136/bmjopen-2025-108346. PMID 41469063